CLINICAL TRIAL: NCT04547881
Title: Prospective Assessment of the Gravity Assisted Technique for Esophageal Endoscopic
Brief Title: Gravity Assisted Technique for Esophageal Endoscopic Submucosal Dissection (ESD)
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Othman, M.D. Chief, Gastroenterology Section, BSLMC William T. Butler Endowed Chair for Distinguished Faculty Associate Professor of Medicine - Gastroenterology and Hepatology Section, Baylor College of Medicine
Other Study IDs: H-44962
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Esophageal Neoplasms
Keywords: Endoscopic Submucosal Dissection; Gravity Assisted Technique
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective data recording study, all patients will receive standard medical care and no experimental interventions will be performed. All patients scheduled to undergo esophageal ESD from December 2018 to December 2021 as medically indicated will be considered for the study, Patients in whom esophageal ESD is considered as part of their standard medical care will be offered to participate in this study. The principle investigator who performing the procedure will also discuss the study with the subjects and ask them to sign a consent. If the patient agrees to participate, he/she will be given the informed consent form and allowed enough time to read it. Then if the patient agrees, he/she will sign the consent form. Data will be prospectively recorded according to the data collection form.

DETAILED DESCRIPTION:
Early precancerous esophageal lesions and esophageal cancer, are a threatening illnesses with high mortality rate, so the early intervention is critical during the course of treatment, statistically, every year an estimated 17,290 adults in the United States will be diagnosed with esophageal cancer. Esophageal cancer is the seventh most common cause of cancer death among men (1, 2). Giving the aggressive nature and fatality of esophageal cancer, the early management using the Endoscopic submucosal dissection is very essential (3).

Esophageal ESD is a technique that grants the en-block resection of lesions, with less morbidity and mortality when compared to surgery, and more efficient than other endoscopic techniques like endoscopic mucosal resection as ESD associated with higher curative resection rates and lower recurrence rates (4). ESD require experience and excellent training due to technique difficulties, longer procedure times and possible serious adverse events.

The esophageal Endoscopic Submucosal Dissection (ESD) is gaining momentum in United States. Although a great deal of training is focused on teaching how to utilize the equipment for performing the procedure, the strategy of where to start the incision and how to proceed with dissection is not yet standardized. The investigators standardized a technique for performing esophageal ESD utilizing gravity as traction to expedite the procedure.

Currently, the investigators are performing this technique for esophageal ESD at Baylor St. Luke's Medical center.

The aim of the study is to assess the mean time needed to perform esophageal ESD using this technique. Our quality metrics are a dissection rate of 9cm2 per hour as suggested by Japanese experts.

Purpose and objective of the study:

1. - Assessing the mean time needed to perform esophageal ESD using this technique. Our quality metrics are a dissection rate of 9cm2 per hour as suggested by Japanese experts.
2. - Assessment of the safety of gravity assisted esophageal ESD.

After obtaining the informed consent, the following information will be collected:

1. - All the incisional times and the submucosal dissection time (details listed below)
2. - Demographic information related to the study participants (age, sex, race, etc.)
3. - BMI
4. - Family History
5. - The pathology reports for ESD.
6. - Social habits such as smoking and drinking alcohol.

The investigator will collect the time that will be spent during this technique as following:

1. - Lower incision time (anal side): this is the initial incision and will start at the anal side of the lesion
2. - Right and left incisional time, these incisions will be on the each side of the lesion and they will meet the initial incision.
3. - The proximal incision time (oral side): is performed at the oral side of the lesion communicating the right and left side incisions.
4. - Total incision time.
5. - Total submucosal dissection time.
6. - Total procedure time

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled to undergo esophageal ESD as part of their standard-of-care.

Exclusion Criteria:

* Patients less than 18 years old.
* Pregnant women
* Patient is unable/unwilling to provide informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled to undergo esophageal ESD from December 2018 to December 2021 as medically indicated will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Total time for lesion removal | 2 years
  To assess the mean time needed to perform esophageal ESD using this technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Cao Y, Liao C, Tan A, Gao Y, Mo Z, Gao F. Meta-analysis of endoscopic submucosal dissection versus endoscopic mucosal resection for tumors of the gastrointestinal tract. Endoscopy. 2009 Sep;41(9):751-7. doi: 10.1055/s-0029-1215053. Epub 2009 Aug 19. PMID 19693750
- See also: Related Info — https://atlas-itn.eu/wp-content/uploads/2020/05/D10-1_main.pdf